CLINICAL TRIAL: NCT02458248
Title: Sodium Intake in Chronic Kidney Disease (STICK): A Randomised Controlled Trial
Brief Title: Sodium Intake in Chronic Kidney Disease (STICK)
Acronym: STICK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College Hospital Galway (Other)
Collaborators: Health Research Board, Ireland (Other); National University of Ireland, Galway, Ireland (Other)
Responsible Party: Principal Investigator, Dr Andrew Smyth, Dr., University College Hospital Galway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRBCRFG-170415-AS
Record Dates: First submitted 2015-05-15; First posted 2015-06-01 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Kidney Diseases; Renal Insufficiency, Chronic; Renal Insufficiency
Keywords: Chronic Kidney Disease; Sodium Reduction; eGFR 30-60ml/min/1.73m2
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium Reduction (Experimental): In addition to usual care, those randomised to the intervention arm will receive specific counseling on behavioural and environmental factors that promote sodium reduction after randomization and at all post-randomisation visits, targeting sodium intake of <100mmol/day (<2.3g/day).
  Interventions: Behavioral: Sodium Reduction
- Usual care (No Intervention): For all participants, standard care will be provided at the nephrology clinic at GUH or by local general practitioners, and includes treatment of hypertension, underlying comorbidities and optimizing the metabolic profile. Participants randomized to usual care will also attend a dietitian-developed healthy eating guidance session but will not receive specific recommendations targeting sodium intake.

INTERVENTIONS:
Behavioral: Sodium Reduction — In addition to usual care, those randomised to the intervention arm will receive specific counseling on behavioural and environmental factors that promote sodium reduction after randomization and at all specified post-randomisation visits, targeting sodium intake of <100mmol/day (<2.3g/day). A research dietitian will develop the specific components of the intervention, based on standardised approaches to education interventions.
  Arms: Sodium Reduction

SUMMARY:
Chronic kidney disease, which affects an estimated 300,000 people in Ireland and over 50 million people in the developed world, is responsible for a considerable burden of premature mortality and morbidity. All patients with chronic kidney disease are recommended low salt diets, i.e. less than a teaspoon of salt per day (which is <5-6g of salt, which contains <2-2.3g of sodium). The average intake in the general population is double the recommended intake, between 1-2 teaspoons per day, which is considered 'moderate' intake. In patients with hypertension, reducing from moderate (average) to low intake is associated with a small reduction in blood pressure. However, achieving this low target salt intake is difficult, and can have a negative knock-on effect on other healthy dietary factors and kidney hormones. In addition, there is no convincing research to show that patients with chronic kidney disease and normal blood pressure benefit from low salt intake. In fact, the small amount of research that does exist shows that the change in kidney function is the same in people who consume low salt diets (<1 teaspoon) and moderate (1-2 teaspoons=average intake) salt diets. Moreover, there are some small studies that report that low-salt diets may increase the risk of death due to heart disease. Given that all patients with chronic kidney impairment are recommended a low-salt diet, it is important that we confirm that this recommendation truly benefits patients. In this randomized controlled trial, we hope to determine whether recommending a low salt intake, compared to average/moderate intake, is associated with a slower rate of decline in kidney function in patients with chronic kidney impairment. The results of this study will provide information to guide future research that will have critical implications for management of patients with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older
* MDRD eGFR of 30-60ml/min/1.73m2 on ≥2 occasions ≥3 months apart
* Most recent eGFR measurement within 3 months Systolic blood pressure <160mmHg and diastolic blood pressure <95mmHg on three office blood pressure readings at time of screening and confirmed by a study ABPM before randomisation of <150/90mmHg
* No change in anti-hypertensive or diuretic medications (including dose) for 3 months before screening visit
* Consumption of moderate sodium intake at screening, defined as an estimated daily sodium intake of >2.3g/day estimated from food frequency questionnaire (FFQ) completed during the screening visit
* Self-reported willingness to modify dietary intake over sustained period, and adhere to directed recommendations over 2 years
* Signed written informed consent

Exclusion Criteria:

* Acute Kidney Injury in the preceding three months, defined as doubling of baseline serum creatinine or rapidly declining eGFR over the preceding six months, defined as a decline in eGFR of ≥10ml/min/1.73m2 in those with established CKD
* Any of the following renal conditions: glomerular disease due to post-infectious glomerulonephritis, IgA nephropathy, thin basement membrane disease, Henoch-Schonlein purpura, proliferative glomerulonephritis, membranous nephropathy (including lupus nephritis), rapidly progressive glomerulonephritis, minimal change disease, or focal segmental glomerulosclerosis
* Prior or planned renal transplantation
* Prior, current or planned renal dialysis
* Medical diagnosis known to be associated with abnormal renal sodium excretion, including Bartter syndrome, SIADH, diabetes insipidus, or serum sodium <125mmol
* Severe heart failure (defined as left ventricular ejection fraction ≤30% or NYHA Class III/IV symptoms)
* High-dose loop or thiazide diuretic therapy, exceeding a total daily dose of frusemide 80mg, bumetanide 2mg, hydrochlorothiazide 50mg, bendroflumethiazide 2.5mg, indapamide 2.5mg, metolazone 2.5mg or the use of both a loop and thiazide diuretic
* Current use of non-steroidal anti-inflammatory drugs (NSAIDs) for 3 or more days per week. Low-dose aspirin <100mg/day is not an exclusion
* Unable to follow educational advice of the research team
* Prescribed high-salt diet, low-salt diet or sodium bicarbonate
* Symptomatic postural hypotension or receiving treatment for postural hypotension
* Current or recent use (within one month) of immunosuppressive medications including tacrolimus, cyclosporine, azathioprine or mycophenolate mofetil
* Pregnancy or lactation
* Unable to comply with 24-hour urinary collections, or medical condition making collection of 24-hour urinary collection difficult (e.g. severe urinary incontinence)
* Participant unlikely to comply with study procedures or follow-up visits due to severe co-morbid illness or other factor (e.g. inability to travel for follow-up visits, drug or alcohol misuse) in opinion of research team
* Cognitive impairment defined as a known diagnosis of dementia, or inability to provide informed consent due to cognitive impairment in the opinion of the investigator
* Body Mass Index (BMI) <20kg/m2 or BMI>40kg/m2
* Participating in another clinical trial or previous allocation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-03; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour urinary creatinine clearance from baseline to final follow-up, measured from 24-hour urinary collection and corresponding serum creatinine measurement at randomisation and final visit. | 24 months

SECONDARY OUTCOMES:
Change in eGFR (MDRD formula) from baseline to final follow-up | 24 months
Change in eGFR (CKD-EPI formula) from baseline to final follow-up | 24 months
Rates of requirement for renal replacement therapy | 24 months
Change in 24-hour urinary protein from baseline to final visit | 24 months
Increase in risk category for prognosis of CKD as measured by the KDIGO 2012 CKD classification table | 24 months
Change in 24-hour urinary sodium excretion from baseline to final visit | 24 months
Change in mean systolic and diastolic blood pressure from 24-hour ambulatory blood pressure monitoring completed at baseline and final visit | 24 months
Composite outcome of change in risk category for prognosis of CKD (increase in risk), requirement for renal replacement therapy or death as measured by the KDIGO 2012 CKD classification table | 24 months
Change in functional status as measured by the assessment functional status questionnaire | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin J O'Donnell, MB PhD MRCPI, Principal Investigator — National University of Ireland, Galway; Andrew Smyth, MB PhD, Principal Investigator — National University of Ireland, Galway
Locations (1):
- HRB Clinical Research Facility Galway, Galway, Ireland

REFERENCES:
- [Derived] Smyth A, Judge C, Kerins C, McDermott S, Niland A, Corcoran C, Dineen R, Alvarez-Iglesias A, Nolan A, Mente A, Griffin MD, O'Shea P, Canavan M, Yusuf S, O'Donnell M. Dietary counselling to reduce moderate sodium intake: effects on cardiovascular and renal biomarkers: primary findings of the COSIP and STICK phase II feasibility randomised controlled trials. EClinicalMedicine. 2023 Feb 15;57:101856. doi: 10.1016/j.eclinm.2023.101856. eCollection 2023 Mar. PMID 37064508
- [Derived] Smyth A, Yusuf S, Kerins C, Corcoran C, Dineen R, Alvarez-Iglesias A, Ferguson J, McDermott S, Hernon O, Ranjan R, Nolan A, Griffin M, O'Shea P, Canavan M, O'Donnell M. Clarifying Optimal Sodium InTake In Cardiovasular and Kidney (COSTICK) Diseases: a study protocol for two randomised controlled trials. HRB Open Res. 2022 Feb 7;4:14. doi: 10.12688/hrbopenres.13210.2. eCollection 2021. PMID 36348660
- [Derived] McMahon EJ, Campbell KL, Bauer JD, Mudge DW, Kelly JT. Altered dietary salt intake for people with chronic kidney disease. Cochrane Database Syst Rev. 2021 Jun 24;6(6):CD010070. doi: 10.1002/14651858.CD010070.pub3. PMID 34164803